CLINICAL TRIAL: NCT03466268
Title: A Phase I Trial to Assess the Safety, Pharmacokinetics, and Anti-tumor Activity of SCC244 in Subjects With Advanced Solid Tumors
Brief Title: Study to Evaluate the Safety and Anti-tumor Activity of SCC244
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Haihe Biopharma Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SCC244-101
Record Dates: First submitted 2017-08-07; First posted 2018-03-15 (Actual); Last update posted 2024-10-09 (Actual); Status verified 2024-03

CONDITIONS: Advanced Solid Tumor
Keywords: Safety; Tolerability; Pharmacokinetics; Anti-tumor activity
MeSH Terms: interventions — glumetinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Dose escalation study of Gumarontinib (Experimental): To determine the maximum tolerated dose (MTD) of Gumarontinib
  Interventions: Drug: Gumarontinib Tablets

INTERVENTIONS:
Drug: Gumarontinib Tablets — Either at 100mgSD、100mgQD、200mgSD、200mgQD、400mgSD、400mgQD、300mgBID、400mgBID
  Other Names: SCC244

SUMMARY:
This study evaluates the Safety, Tolerability, Pharmacokinetics, and Anti-tumor Activity of SCC244 in patients with advanced solid tumors with c-Met Alterations.

DETAILED DESCRIPTION:
A Phase I Dose Escalation and Dose Expansion Trial to Evaluate the Safety, Pharmacokinetics and Anti-tumor Activity of SCC244, a Highly Selective c-Met Inhibitor, in Patients with Advanced Non-small Cell Lung Cancer.

Phase Ia: The primary objective is to determine the MTD, BED and recommended dose for Phase Ib in patients with advanced NSCLCs. In addition, the safety, tolerability, preliminary efficacy and PK of SCC244 and its metabolites will also be evaluated. In phase Ia, planned dose levels will be evaluated with a starting dose of 100mg.

Phase Ib: The primary objective is to assess the ORR in advanced NSCLC patients with c-MET change. The DOR, DCR, TTR, PFS, one-year OS rate, safety, tolerability, and PK will also be evaluation in Phase Ib.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subject ≥ 18 years of age.
2. Life expectancy ≥ 12 weeks by the Investigator.
3. In Phase Ia, histologically confirmed NSCLC (including sarcomatoid carcinoma) with c-Met alterations defined as c-Met gene amplification ≥ 5 copies or c-Met protein overexpression (IHC 3+) or c-Met exon 14 skipping mutation. No EGFR T790M mutation for subjects with c-Met gene amplification or c-Met protein overexpression; KRAS/ALK/ROS1 WT or unknown mutation/rearrangement status for subjects with c-Met exon 14 skipping mutation.
4. In Phase Ib, histologically confirmed NSCLC as in Phase Ia, AGC, or HCC with c-Met gene amplification ≥ 5 copies, or c-Met protein overexpression (IHC 3+). HCC subjects must have Child Pugh Class A.
5. Available fresh samples of NSCLC (except for c-Met exon 14 skipping mutation that can be from archival tumor sample), and available fresh or archival tumor sample of AGC and HCC for c-Met gene alteration characterization or determination of c-Met protein overexpression (IHC 3+). Fine needle aspiration and cytology samples are not sufficient.
6. In Phase Ia/Ib, all NSCLC subjects with EGFR mutation must have progressive disease after 1 or 2 lines of prior therapy including at least an EGFR-TKI targeting other than c-Met alterations. Subjects with c-Met exon 14 skipping mutation must have received at least 1 line of standard therapy in Phase Ia and can be first or second line subjects in Phase Ib. In Phase Ib, subjects with AGC must have progressive disease after at least 1 line of prior standard therapy and subjects with HCC must have received 1 line of targeted agent therapy.
7. At least 1 measurable target lesion.
8. Eastern Cooperative Oncology Group (ECOG) performance score 0-2.
9. Adequate organ function as documented
10. Toxicities from any prior therapy, surgery, or radiotherapy must have resolved to Grade 0 or 1 as per the National Cancer Institute- Common Terminology Criteria for Adverse Events (NCI-CTCAE), excluding alopecia.

Exclusion Criteria:

1. Pregnant (serum human chorionic gonadotropin positive) or breastfeeding female subject.
2. Prior anti-tumor systemic chemotherapy or loco-regional therapy for HCC (such as percutaneous ethanol injection, chemoembolization or radiofrequency ablation), biologics therapy, Chinese herbal anti-cancer or anti-infective medication within 28 days or 5 × half life time, whichever occurs last, before the first dose.
3. Prior therapy with another c-Met inhibitor.
4. Presence of EGFR T790M mutation in NSCLC subjects pretreated with an EGFR-TKI; Known KRAS/ALK/ROS1 mutation/rearrangement in NSCLC subjects with c-Met exon 14 skipping mutation.
5. Known or suspected hypersensitivity to SCC244 and/or its excipients.
6. Palliative radiotherapy to bone metastasis within 4 weeks prior to the first dosing.
7. Prior or concomitant other malignant tumor (except effectively controlled non-melanoma skin cancer, breast carcinoma in situ or cervix cancer in situ and superficial bladder cancer within past 5 years).
8. Cardiac function impairment or clinically significant heart disease including congestive heart-failure ≥ Grade 2 according to grading of New York Heart Association, arrhythmia, conduction abnormality requiring treatment, myocardium diseases or uncontrollable hypertension within 6 months prior to screening. QTc-prolongation > 470 msec, risk factors for Torsades De Pointe, hypokalemia or family history of long-QT-Syndrome.
9. History of stroke within 6 months prior to screening.
10. Known central nervous system or brain metastasis that is either symptomatic or untreated. Metastases that have been treated by complete resection and/or radiotherapy demonstrating stability or improvement are not an exclusion criterion provided they are stable as shown by CT scan for at least 1 month without evidence of cerebral edema and no requirements for corticosteroids or anticonvulsants.
11. Inability to swallow oral medication, or active digestive system disease, or major digestive surgery, which in the Investigator's opinion can affect administration and absorption of SCC244 (such as active ulcerative disease, uncontrollable diarrhea, and small bowel resection).
12. Any disease or condition with clinical significance (such as pancreatitis, uncontrollable diabetes, active or uncontrollable infection, drug or alcohol abuse, or psychiatric conditions), which can affect protocol compliance.
13. Positive result for active infection by hepatitis B or C virus (HBV or HCV); known positivity for human immunodeficiency virus (HIV) infection.
14. Men and women of reproductive potential not willing or not able to employ a highly effective method of birth control/contraception to prevent pregnancy until the end of trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2017-09-14 (Actual); Primary Completion 2023-01-09 (Actual); Study Completion 2023-01-09 (Actual)

PRIMARY OUTCOMES:
DLT(Dose limit toxity) | 35 days
  To evaluate the DLT in patients with advanced solid tumor
MTD(Max tolerance does) | 35 days
  To evaluate the MTD in patients with advanced solid tumor
BED(Biological effective dose) | 35 days
  To evaluate the BED in patients with advanced solid tumor
ORR(Objective response rate) | 8 weeks
  To evaluate the ORR in patients with advanced solid tumor in Ib

CONTACTS AND LOCATIONS:
Overall Officials: Yilong Wu, M.D., Principal Investigator — Guangdong Provincial People's Hospital
Locations (1):
- Guangdong General Hospital, Guangzhou, Guangzhou, China